CLINICAL TRIAL: NCT02940314
Title: A Randomized, Open-label, Single Dose, 2-way Crossover Study to Compare the Safety and Pharmacokinetic Characteristics After Administration of HIP1503 and HGP1103 in Healthy Male Volunteers
Brief Title: Safety and Pharmacokinetic Characteristics After Administration of HIP1503 and HGP1103 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-SOLT-101
Record Dates: First submitted 2016-10-19; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sequence 1 (Experimental): HGP1103→HIP1503
  Interventions: Drug: HIP1503; Drug: HGP1103
- Sequence 2 (Experimental): HIP1503→HGP1103
  Interventions: Drug: HIP1503; Drug: HGP1103

INTERVENTIONS:
Drug: HIP1503
  Other Names: Solifenacin tartrate 10.66 mg
Drug: HGP1103
  Other Names: Solifenacin succinate 10 mg

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetic characteristics after administration of HIP1503 and HGP1103 in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age 19 to 45 years.
2. The result of Body Mass Index(BMI) 17.5 kg/m2~ 30.5 kg/m2, body weight over 55kg.
3. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing.

Exclusion Criteria:

1. Presence of medical history or a concurrent disease, including clinically significant disorders in kidney, liver, cardiovascular system, respiratory system, endocrine system, or neuropsychiatric system.
2. Medical history of Gastrointestinal Diseases that effects drug absorption (esophageal disease, chronic disease) or surgery( except appendectomy , herniolaparotomy)
3. sit SBP > 140 mmHg, sit DBP > 90 mmHg
4. Alcohol or Drug abuse within 1 year

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
AUClast | 0h(Predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72hours (total 14)
Solifenacin Cmax | 0h(Predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72hours (total 14)

SECONDARY OUTCOMES:
Solifenacin AUCinf | 0h(Predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72hours (total 14)
Solifenacin Tmax | 0h(Predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72hours (total 14)
Solifenacin t1/2 | 0h(Predose), 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72hours (total 14)

IPD SHARING:
Plan to Share IPD: No